CLINICAL TRIAL: NCT03485157
Title: A Phase 2B, Prospective, Double-blinded, Randomized Controlled Trial of the Micronized Dehydrated Human Amnion Chorion Membrane Injection as Compared to Saline Placebo Injection in the Treatment of Osteoarthritis of the Knee
Brief Title: Micronized dHACM vs. Saline in the Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIOA001
Record Dates: First submitted 2018-03-20; First posted 2018-04-02 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Micronized dHACM (Experimental): Injection of micronized dHACM
  Interventions: Biological: Micronized dHACM
- Saline (Placebo Comparator): Injection of 0.9% Sodium Chloride Injection, USP
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Micronized dHACM — Injection of 40 mg micronized dehydrated human amnion chorion membrane (dHACM) suspended in 1 mL 0.9% Sodium Chloride, USP
  Arms: Micronized dHACM
Drug: Saline — Injection of 1 mL 0.9% Sodium Chloride, USP
  Arms: Saline

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of micronized dehydrated human amnion chorion membrane as compared to the 0.9% Sodium Chloride Injection, USP placebo control for the treatment of knee osteoarthritis

DETAILED DESCRIPTION:
Each subject will receive 1 injection (micronized dHACM or placebo) and be evaluated for efficacy and safety during a 12-month observation period. A second injection (open-label access to micronized dHACM) will be offered to all subjects at the 180-day, 270-day, and 365-day time points, it may only be used once. Blinding for the first injection treatment allocation will be maintained until the end of the study.

Subjects who receive the open-label access treatment will continue to be followed for 180 days after this second injection, regardless of the time at which treatment was received.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 and ≤ 80 years
2. Subject has a diagnosis of osteoarthritis (OA) defined as Grade 1 to 3 on the Kellgren Lawrence grading scale
3. Subject is willing and able provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study
4. Subject must have a VAS pain scale greater than 45

Exclusion Criteria:

1. Subject has a diagnosis of osteoarthritis (OA) defined as Grade 4 on the Kellgren Lawrence grading scale
2. BMI greater than 40 kg/m^2
3. Subject has active infection at the injection site
4. Symptomatic OA of the contralateral knee or of either hip that is not responsive to acetaminophen (Tylenol®) and requires other therapy.
5. Subject has rheumatoid arthritis, psoriatic arthritis, or have been diagnosed with any other disorders that is the primary source of their knee pain, including but not limited to: osteonecrosis, radiculopathy, bursitis, tendinitis, tumor, cancer
6. Subject has documented history of gout or pseudo-gout
7. Subject has autoimmune disease or a known history of having Acquired Immunodeficiency Syndromes (AIDS) or HIV
8. Subject has received any of the following to the target knee:

   1. Intra-articular hyaluronic acid (HA) injection within 12 weeks prior to screening
   2. Steroid or platelet rich plasma (PRP) injection within 12 weeks prior to screening
   3. Has had or is planning to have major surgery or arthroscopy in the target knee within 26 weeks of treatment
   4. History of a total knee arthroplasty
9. Subject has used an investigational drug, device or biologic within 12 weeks prior to treatment
10. Subject has a history of immunosuppressive or chemotherapy in the last 5 years
11. Subject has had prior radiation at the site
12. Subject is currently taking anticoagulant therapy (excluding Plavix or Aspirin)
13. Subject is pregnant or plans to become pregnant within 365 days of treatment
14. Subject has any significant medical condition that, in the opinion of the Investigator, would interfere with protocol evaluation and participation
15. Subject is a worker's compensation patient
16. Subject is a prisoner

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred C Gellhorn, MD, Principal Investigator — Esprit R&D Associate GSK
Locations (17):
- United States (17):
  - Central Research Associates, Inc, Birmingham, Alabama
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Horizon Clinical Research, La Mesa, California
  - UConn Health, Farmington, Connecticut
  - Bone & Joint Inst. at Hartford Hospital, Hartford, Connecticut
  - Gulfcoast Research Institute, Sarasota, Florida
  - Paragon Sports Medicine, Atlanta, Georgia
  - Hinsdale Orthopedics, Hinsdale, Illinois
  - Arthritis Care Specialist of Maryland, Columbia, Maryland
  - MedSport, Ann Arbor, Michigan
  - Weill Cornell Medicine, New York, New York
  - Wake Reseach, Durham, North Carolina
  - Wake Research, Raleigh, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - SAMMC, Fort Sam Houston, Texas
  - Ortho Virginia, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening visit occurred after enrollment and could possibly be the same day as randomization/treatment.
Period: Double Blind Phase
Arm/Group | Micronized dHACM | Saline
Started | 223 | 224
Completed | 208 | 203
Not Completed | 15 | 21
Not completed — Lost to Follow-up | 4 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Removal by PI | 3 | 7
Period: Open Label Phase
Arm/Group | Micronized dHACM | Saline
Started | 108 | 109
Completed | 104 | 104
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Removal by PI | 2 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics of subjects in the ITT Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Micronized dHACM | Saline | Total
Number analyzed (Participants) | 223 | 224 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.89 (10.619) | 58.45 (11.294) | 58.17 (10.954)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 140 | 260
  Male | 103 | 84 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 211 | 212 | 423
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 24 | 19 | 43
  White | 193 | 195 | 388
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Height (in) [Mean (Standard Deviation); unit: Inches] | 67.17 (4.114) | 66.72 (3.748) | 66.94 (3.937)
Weight [Mean (Standard Deviation); unit: lbs] | 187.22 (39.629) | 185.12 (40.305) | 186.17 (39.938)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.74 (4.919) | 29.81 (5.279) | 29.77 (5.097)

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: Change From Baseline in Visual Analog Scale (VAS) for Pain at 90 Days
Description: Visual Analog Scale (VAS): 0 to 100 mm horizontal visual analog scale with a higher score indicating greater pain
Time Frame: 90 days
Population: Population: Intent To Treat Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Micronized dHACM | Saline
Number analyzed (Participants) | 223 | 224
score on a scale
  Value | 32.8 (26.39) | 34.1 (26.40)
  Change from baseline | -35.1 (26.72) | -34.2 (26.87)

2. Primary Outcome: Primary Efficacy Endpoint: Change From Baseline in Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index at 90 Days
Description: Western Ontario and McMaster Universities Arthritis Index (WOMAC) evaluation of Hip and Knee Osteoarthritis. Self-administered questionnaire consisting of 24 questions divided into 3 subscales:
  * Pain (5 questions)
  * Stiffness (2 questions)
  * Physical Function (17 questions)
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score, with a possible total score range of 0-96.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: 90 days
Population: Population: Intent To Treat Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Micronized dHACM | Saline
Number analyzed (Participants) | 223 | 224
score on a scale
  Value | 26.9 (18.43) | 28.8 (18.98)
  Change from baseline | -20.6 (18.16) | -19.6 (17.99)

3. Primary Outcome: Primary Safety Endpoint: Number of Participants With Adverse Events (AEs)
Description: Number of Participants with At Least 1 Treatment Emergent Adverse Event (TEAE) Reported
Time Frame: 365 days
Population: Subjects with at least 1 Treatment Emergent Adverse Event reported
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized dHACM | Saline
Number analyzed (Participants) | 223 | 224
Participants | 123 | 120

4. Primary Outcome: Primary Safety Endpoint: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of Participants with At Least 1 Serious Treatment Emergent Adverse Event (TEAE) Reported
Time Frame: 365 days
Population: Subjects reporting Serious Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized dHACM | Saline
Number analyzed (Participants) | 223 | 224
Participants | 11 | 12

5. Primary Outcome: Primary Safety Endpoint: Number of Participants With Unanticipated Adverse Events
Description: Number of Participants with At Least 1 Unanticipated Treatment Emergent Adverse Event (TEAE) Reported
Time Frame: 365 days
Population: Subjects reporting Unanticipated Treatment Emergent Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized dHACM | Saline
Number analyzed (Participants) | 223 | 224
Participants | 16 | 16

6. Secondary Outcome: Secondary Endpoint: Change From Baseline in Visual Analog Scale (VAS) at 180 Days
Description: Visual Analog Scale (VAS) : 0 to 100 mm horizontal visual analog scale with a higher score indicating greater pain
Time Frame: 180 days
Population: Population: Intent To Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Micronized dHACM | Saline
Number analyzed (Participants) | 223 | 224
score on a scale
  Value | 31.1 (26.98) | 32.2 (27.35)
  Change From Baseline | -36.9 (28.51) | -36.1 (27.94)

7. Secondary Outcome: Secondary Endpoint:Change From Baseline in WOMAC at 180 Days
Description: as for outcome 2
Time Frame: 180 days
Population: Population: Intent To Treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Micronized dHACM | Saline
Number analyzed (Participants) | 223 | 224
score on a scale
  Value | 26.0 (19.45) | 27.6 (19.63)
  Change From Baseline | -21.6 (20.91) | -20.8 (20.67)

8. Other Pre Specified Outcome: Exploratory Endpoint: Change From Baseline in the Visual Analog Scale (VAS) for Pain at 270, and 365 Days
Description: VAS: 0 to 100 mm horizontal visual analog scale with a higher score indicating greater pain
Time Frame: Up to 365 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory Endpoint: Change From Baseline in the WOMAC Scores at 270 and 365 Days
Description: as for outcome 2
Time Frame: Up to 365 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory Endpoint: Change From Baseline in the Visual Analog Scale (VAS) for Satisfaction at 90, 180, 270 and 365 Days
Description: VAS: 0 to 100 mm horizontal visual analog scale with a higher score indicating greater satisfaction
Time Frame: Up to 365 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory Endpoint: Change From Baseline in the KOOS Scores at 90, 180, 270, and 365 Days
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS): 5 subscales scored on a 5 point scale where the final score is summed and transformed into a 100 point scale with a higher score representing no disability and a lower score representing extreme disability
Time Frame: Up to 365 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collects for 1 year in the double blinded study and 6 months in the Open Label Study.
Groups:
- Open-Label Micronized dHACM: Open-label injection of micronized dHACM
  Micronized dHACM: Injection of 40 mg micronized dehydrated human amnion chorion membrane (dHACM) suspended in 1 mL 0.9% Sodium Chloride, USP
Arm/Group | Micronized dHACM | Saline | Open-Label Micronized dHACM
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/224 | 0/217
Serious Adverse Events (participants affected / at risk) | 11/223 | 12/224 | 5/217
Other Adverse Events (participants affected / at risk) | 123/223 | 120/224 | 94/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micronized dHACM (N=223) | Saline (N=224) | Open-Label Micronized dHACM (N=217)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Injection site joint pain (General disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micronized dHACM (N=223) | Saline (N=224) | Open-Label Micronized dHACM (N=217)
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 49 | 29
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 11 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 8 | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 10 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Joint noise (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthroplasty (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Injection site joint pain (General disorders) | 14 | 2 | 21
Oedema peripheral (General disorders) | 7 | 2 | 3
Injection site joint swelling (General disorders) | 3 | 0 | 9
Injection site oedema (General disorders) | 2 | 1 | 0
Injection site pain (General disorders) | 1 | 2 | 1
Pain (General disorders) | 0 | 2 | 1
Peripheral swelling (General disorders) | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Effusion (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0
Injection site mass (General disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 2
Injection site swelling (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 5 | 4
Muscle strain (Injury, poisoning and procedural complications) | 1 | 4 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 2 | 5
Joint injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 3 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 0
Sinusitis (Infections and infestations) | 2 | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 1
Latent syphilis (Infections and infestations) | 0 | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral respiratory infection (Infections and infestations) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Restless leg syndrome (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Mouth swelling (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 2 | 2 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 2 | 3
Thyroid hormones increased (Investigations) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Veritgo (Ear and labyrinth disorders) | 3 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1 | 0
Foot operation (Surgical and medical procedures) | 1 | 0 | 0
Knee arthoroplasty (Surgical and medical procedures) | 1 | 0 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Post cholecystectomy hyperplasia (Hepatobiliary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Injection site discomfort (General disorders) | 0 | 0 | 1
Injection site joint movement impairment (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1
Immunisation reaction (Immune system disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/57/NCT03485157/Prot_004.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT03485157/SAP_005.pdf